CLINICAL TRIAL: NCT01374334
Title: Lower Extremities Muscle Strength and Power Thresholds Required for Mobility Independence in Older Adults
Brief Title: Lower Extremities Muscle Strength and Power Thresholds Required for Mobility Independence
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Moshe Marko, Assistant professor
Other Study IDs: ThresholdMarko
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2010-08

CONDITIONS: Physical Disability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Aging is associated with loss of muscle strength and a serious import of physical disability. Treatment of age-related physical disability should focus on the prevention of the condition rather than the consequences. Need to modify daily tasks is an early sign of future mobility disability. Many older adults who utilize daily task modifications report no mobility difficulty. Neglect to self-report task modification may delay intervention. Identifying objective marker of task modification will help to identify task modifiers.

DETAILED DESCRIPTION:
Background: There is a significant rise in the number of people who are living well into old age. Aging is associated with loss of muscle strength and a serious import of physical disability. Age-related physical disability is associated with physical dependence, poor quality of life, and mortality. Treatment of age-related physical disability should focus on the prevention of the condition rather than the consequences. Need to modify daily tasks is an early sign of future mobility disability. Many older adults who utilize daily task modifications report no mobility difficulty. Neglect to self-report task modification may delay intervention. Identifying objective marker of task modification will help to identify task modifiers. Loss of muscle strength is associated with mobility decline. Older adults who engage in habitual physical activity (PA) are more likely to maintain physical independence until shortly before the natural end of their lives. Yet, many older adults are not physically active. Health-care professional in general and physical therapists in particular, are in a unique position to promote PA among older adults. Healthcare providers who habitually engage in PA are more likely to consult their patients on PA guidelines.

Purposes: The purposes of the following studies were to: 1) examine lower extremity muscle strength across subjects who do, and do not utilize task modifications, 2) to determine the strength of the association between lower extremity muscle strength and daily task modifications in older adults living independently, 3) identify functionally relevant isometric and isokinetic cutpoints of lower extremity muscle strength below which daily task modifications are more prevalent, 4) to compare the relative diagnostic accuracy of isometric versus isokinetic strength cutpoints as they relate to daily task modifications, 5) estimate the rate of participation in moderate and vigorous physical activity (PA) among student physical therapists (SPTs), 6) compare these estimates to rates of PA among US adults, and 7) assess barriers to PA among SPTs

Methods: To address the first two purposes, fifty-three community dwelling male (21) and female (32) older adults (76.4±5.2 years) were observed performing a chair rise, negotiating stairs, kneeling from a standing position, and rising from supine to stand. Levels of daily task modifications were assessed using a previously described, valid, and reliable tool [MOD]. The MOD assesses task modifications using six hierarchically ranked categories from zero (no modification) to five (refusal). Rankings were summed across tasks. A score of ≥5 points on the summed MOD score was the cutpoint between a classification of daily Task-Modifiers (TM) and None-Task-Modifiers (NTM). Normalized to body weight Isometric measures of peak muscle torque were obtained from the hip extensors, knee extensors, and ankle plantar flexors using a Biodex testing device. A net anti-gravity composite measure of isometric lower extremity muscle force production in the sagittal plane (NETforce) was calculated by summing the normalized torques from the three muscle groups. An independent t-test was used to compare groups (TM vs. NTM) across the dependent measures of muscular torque. A logistic regression model was used to determine the association between torque measures and group assignment.

To address the third and the forth purposes same fifty-three community dwelling male (21) and female (32) older adults (76.4±5.2 years) were observed performing same activities as above. Normalized to body weight isometric and isokinetic (60⁰ per second) measures of peak muscle strength were obtained from the hip extensors, knee extensors, and ankle plantar flexors using a Biodex Isokinetic testing device. A composite torque outputs were calculated by summing the normalized torques from the three muscle groups. An independent t-test was used to compare groups (TM vs. NTM) across the dependent measures of muscular torque. Discriminant analysis{{1397 Hasegawa,R. 2008}} was repeated for each predictor variable separately to determine the minimal strength cutpoints of normalized composite lower extremity isometric and isokinetic strength outputs that would optimally differentiate between the TM and NTM groups. An ROC curve analysis was performed to determine the sensitivity and specificity. A repeated, separated logistic regression with the group classification as the dependent variable and the lower extremity strength measures as the independent variables was conducted. For all statistical tests, a P-value of less than 0.05 was considered statistically significant. All data analyses were performed using SPSS (version 18; SPSS Inc., Chicago, IL, USA). A p value of .05 was used the reject the null hypothesis.

To address the last three purposes, we applied a cross-sectional survey design [N = 126 SPTs enrolled in a professional (entry level) physical therapist education program]. Frequencies, percentages, and cross-tabulations followed by chi-square tests were used to address purposes number 5 and 6. Qualitative (coding) followed by non-parametric statistical procedures were used to assess purpose number 7.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* no major health problems

Exclusion Criteria:

* Participants were not invited for further testing if they were unable to understand basic English, or reported health problems that contraindicated strength and functional testing.
* Examples of such exclusion criteria included severe orthopedic limitations, uncontrolled cardiovascular or metabolic diseases, recent/unhealed fractures, disorders with highly variable course (e.g. multiple sclerosis), severe cognitive impairments, or a score of 20/30 or below on the Mini-Mental State Examination (MMSE) test (Folstein,M.F. 1975; Jensen,J. 2003;Tombaugh,T.N. 1992;).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: fifty-three community dwelling male (21) and female (32) older adults (76.4±5.2 years) were observed performing a chair rise, negotiating stairs, kneeling from a standing position, and rising from supine to stand.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Marko, Principal Investigator — State University of New York - Upstate Medical University